CLINICAL TRIAL: NCT01542008
Title: Treatment Adherence Enhancement in Bipolar Disorder
Acronym: CAE RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor of Psychiatry, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH0933 21-01A1; 1R01MH0933 21-01A1 (Other Grant/Funding Number: National Institite of Mental Health)
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Treatment Noncompliance; Bipolar Disorder
MeSH Terms: conditions — Patient Compliance; Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Customized Adherence Enhancement (CAE) (Experimental): This arm will receive the CAE intervention.
  Interventions: Behavioral: Customized Adherence Enhancement (CAE)
- broad non-individualized education (EDU) (Active Comparator): This arm will receive the EDU intervention.
  Interventions: Behavioral: broadly-directed, non-individualized education (EDU)

INTERVENTIONS:
Behavioral: Customized Adherence Enhancement (CAE) — CAE consists of the application of a series of up to four psychosocial treatment modules based upon a baseline evaluation of adherence vulnerabilities/needs. The standardized modules (Psychoeducation, Modified Motivational Enhancement Therapy, Communication with Providers, Medication Routines), are assigned based upon pre-established criteria designed to fit the needs of the patient.
  Arms: Customized Adherence Enhancement (CAE)
Behavioral: broadly-directed, non-individualized education (EDU) — EDU will consist of 4 core in-person sessions using the patient work-book from the NIMH funded study, Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD), and following the general educational format of the Collaborative Care "control" intervention in the STEP study. EDU addresses BD treatment broadly, including diagnosis and management, and the sessions will review the materials and allow time for questions as needed.
  Arms: broad non-individualized education (EDU)

SUMMARY:
Bipolar disorder (BD) is a serious and chronic mental illness that is associated with substantial impairment in quality of life and functional outcomes, high rates of suicide, and high financial costs. In spite of a proliferation of treatments for BD, nearly half of individuals with BD do not benefit from pharmacotherapy because of sub-optimal medication treatment adherence. Non-adherence with BD medication treatment dramatically worsens outcomes. Reasons for non-adherence among individuals with BD are multi-dimensional, and it has been suggested that adherence enhancement might work best if the intervention specifically addresses factors that are important and modifiable for a specific individual. In spite of the enormity of the problem, the literature on interventions to improve treatment adherence is surprisingly limited. There is an urgent need for interventions to enhance treatment adherence among BD patients that: 1) are at high risk for future treatment non-adherence; 2) may not have access to or interest in long-term, high-intensity, and specialized care; and 3) are flexible and patient-focused taking into account reasons for non-adherence for a specific individual.

The proposed study is a first-ever RCT focused specifically on BD treatment adherence enhancement, and will test whether a customized adherence enhancement (CAE) psychosocial intervention improves adherence and mental health outcomes compared to broadly-directed, non-individualized education (EDU). The proposed project has the potential to greatly advance the care of BD patients who are at greatest risk for poor health outcomes, with findings expected to be generalizable across a variety of treatment settings.

Hypothesis 1: CAE will be associated with greater improvement in treatment adherence compared to broadly-directed, non-individualized BD education (EDU).

Hypothesis 2: CAE will be associated with improved BD symptoms compared to EDU.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have type I or type II Bipolar Disorder (BD) as confirmed by the Structured Clinical Interview for DSM-IV Axis I Disorders Patient Version (SCID-P)
* Have had BD for at least two years duration
* Have received treatment with at least one evidence-based medication to stabilize mood for at least six months (lithium, anticonvulsant, or antipsychotic mood stabilizer)
* Either 20% or more non-adherent with current BD medication treatment (i.e. lithium, anticonvulsant, or antipsychotic mood stabilizer)

Exclusion Criteria:

* Unable or unwilling to participate in psychiatric interviews. This will include individuals, who may be too psychotic to participate in interviews/rating scales
* Unable or unwilling to give written, informed consent to study participation
* Individuals at high risk for suicide who can not be safely managed in their current treatment setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2012-04; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Tablet Routine Questionaire (TRQ) "past month" item at 24 weeks | Baseline and 24 weeks
  The TRQ "past month" item is a subject report of the percentage of prescribed medications not taken within the past month.
Change from baseline in the Tablet Routine Questionaire (TRQ) "past week" item at 24 weeks | Baseline and 24 weeks
  The TRQ "past week" item is a subject report of the percentage of prescribed medications not taken within the past week.
Change from baseline in treatment adherence as measured by special pill cap counter at 24 weeks | Baseline and 24 weeks
  A special pill cap will record the time/date of bottle opening. The cap will be used for the medication that the patient takes the most frequently (in the case of multiple BD medications taken at same frequency, the medication that was started most recently will be selected). A dose will be counted as "taken" if the bottle is opened within two hours of the prescribed time. A percent of doses taken (treatment adherence) will be calculated by dividing the number of times the bottle is opened by the number of times it should have been opened as per the prescription.

SECONDARY OUTCOMES:
Change from baseline in Brief Psychiatry Symptom Scale (BPRS) at 24 weeks | baseline and 24 weeks
Change from baseline in Montgomery Asberg Depression Rating Scale (MADRS) at 24 weeks | baseline and 24 weeks
Change from baseline in Young Mania Rating Scale (YMRS) at 24 weeks | baseline and 24 weeks
Change from baseline in Clinical Global Impression, Bipolar Version (CGI-BP) at 24 weeks | baseline and 24 weeks
Change from baseline in Global Assessment of Functioning (GAF) at 24 weeks | baseline and 24 weeks
Change from baseline in General Self Efficacy Scale at 24 weeks | baseline and 24 weeks
Change from baseline in the Drug and Alcohol portion of the Addiction Severity Index (ASI) at 24 weeks | baseline and 24 weeks
Change from baseline in Treatment alliance (Trust in Providers scale) at 24 weeks | baseline and 24 weeks
Change from baseline in Stigma for Mental Illness Scale at 24 weeks | baseline and 24 weeks
Change from baseline in Drug Attitudes Inventory (DAI) at 24 weeks | baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Aftab A, Levin J, Aebi M, Bhat C, Sajatovic M. Associations of Comorbid Anxiety With Medication Adherence and Psychiatric Symptomatology in a Population of Nonadherent Bipolar Disorder Subjects. J Nerv Ment Dis. 2018 Apr;206(4):258-262. doi: 10.1097/NMD.0000000000000788. PMID 29351117